CLINICAL TRIAL: NCT04533230
Title: Prevention of Benzodiazepine Misuse: A Randomized Trial in Primary Care
Brief Title: Prevention of Benzodiazepine Misuse in Primary Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to the COVID-19 pandemic restricting access to primary healthcare clinics.
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Franck, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1347-31/2
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Benzodiazepine Dependence; Benzodiazepine Abuse; Substance Use Disorders
Keywords: Primary Health Care; Benzodiazepines; Substance Use Disorder; Addiction; Prescription Drugs
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Karolinska Trial Alliance (KTA) will conduct the randomization. The administrator at KTA who conducts the randomization will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Educational intervention with prescription feedback (Experimental): The manager and physicians at each intervention center will participate in a brief educational intervention about benzodiazepines and benzodiazepine-like hypnotics and receive 12 months of targeted feedback on prescription of these drugs. The education will cover national and regional treatment guidelines for anxiety, depression, and insomnia, which include guidelines on prescription of benzodiazepines and benzodiazepine-like hypnotics.
  Interventions: Behavioral: Educational intervention with prescription feedback
- Information on guidelines (Active Comparator): The manager and physicians at each center in the active control group will receive written information on national and regional treatment guidelines for anxiety, depression, and insomnia, which include guidelines on prescription of benzodiazepines and benzodiazepine-like hypnotics. These centers will not receive the onsite educational intervention or 12 months of targeted prescription feedback.
  Interventions: Behavioral: Information on treatment guidelines
- No active intervention: standard care (No Intervention): The manager and physicians at each primary health care center in the passive control group will receive no active intervention. The passive control group will consist of primary health care centers that are not actively participating in the study. Data will be gathered from regional registers and databases. Thus, there will be no need to contact or communicate directly with the centers. This arm will be used only if the General Data Protection Regulation continues to allow access to regional registers and databases in primary health care.

INTERVENTIONS:
Behavioral: Educational intervention with prescription feedback — Educational intervention and targeted feedback on prescription of benzodiazepines and benzodiazepine-like hypnotics
  Arms: Educational intervention with prescription feedback
Behavioral: Information on treatment guidelines — Written information on treatment guidelines.
  Arms: Information on guidelines

SUMMARY:
Benzodiazepines and benzodiazepine-like hypnotics (z-drugs) are prevalent and addictive narcotics. Guidelines recommend restricted prescription of these drugs for anxiety and insomnia. The majority of benzodiazepine prescriptions are written for these disorders by physicians (GPs) in primary health care. Primary health care is thus an important arena for efforts to reduce access to benzodiazepines in order to lower the number of new users and users at risk of dependency. This trial evaluates whether a brief educational intervention in primary health care followed by 12 months of feedback on prescription data changes the prescription of benzodiazepines and benzodiazepine-like hypnotics.

DETAILED DESCRIPTION:
Background: Benzodiazepines and the benzodiazepine-like hypnotics, often called "z-drugs" (hereafter "benzodiazepines") are common and addictive narcotic drugs that can be obtained by prescription. Even short-term prescription can become a long-term problem, leading to tolerance and dependency, as well as adverse effects, including cognitive disturbance and decline, behavioral problems, emergency visits, accidents, suicide, and drug-related mortality. Guidelines restrict prescription of these drugs for anxiety and insomnia. The majority of benzodiazepine prescriptions are written for these disorders by physicians in primary health care. Primary health care is thus an important arena for efforts to reduce access to benzodiazepines in order to lower the number of new users and users at risk of dependency.

Aim: This randomized controlled trial tests whether a brief educational intervention in primary health care followed by 12 months of feedback on prescription data changes prescriptions of benzodiazepines and benzodiazepine-like hypnotics.

Methods: Primary health care centers will be invited to participate in the study. Centers that express interest in participating, meet the inclusion criteria, and do not meet the exclusion criteria will be randomized to the intervention or the control group. Personnel at the intervention centers will participate in a brief educational intervention followed by 12 months of regular feedback on benzodiazepine prescriptions that are written at the center. Personnel in an active control group will receive written information on treatment guidelines but will not receive the onsite educational intervention or prescription feedback. Data on characteristics of participating primary health care centers, as well as on prescriptions before the intervention and during and after the 12-month follow-up period, will be gathered from regional health care registers and databases and statistically analyzed.

ELIGIBILITY:
Inclusion criteria for primary health care centers:

* Employs at least two full-time physicians
* Has at least 3000 patients
* Has a regional care agreement (contract)

Exclusion criteria for primary health care centers:

* In operation for less than 12 months
* Participated in an intervention to reduce benzodiazepine prescriptions in the last 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prescriptions of benzodiazepines and benzodizepine-like hypnotics | 12 months
  Change in total prescriptions

SECONDARY OUTCOMES:
New prescriptions of benzodiazepines and benzodiazepine-like hypnotics | 12 months
  Change in new prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Johan Franck, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Region Stockholm, Academic primary health care center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data for this study will be gathered from regional registers and health care databases. For permission to access these data, interested parties should contact the regions.
Supporting Information: Study Protocol
Time Frame: Interested parties can contact the regions to request data from regional registers and databases.
Access Criteria: Access criteria for data sharing are determined by the regions and regulated by law.
URL: https://skr.se/